CLINICAL TRIAL: NCT01953770
Title: Moscow-Berlin 2008 Multicenter Randomised Study for Treatment of Acute Lymphoblastic Leukemia in Children and Adolescents
Brief Title: Childhood Acute Lymphoblastic Leukemia Treatment Protocol Moscow-Berlin 2008
Acronym: ALL-MB 2008
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Principal Investigator, Karachunskiy Alexander, Deputy director of Research Institute of Pediatric Hematology, Oncology and Immunology, Federal Research Institute of Pediatric Hematology, Oncology and Immunology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALL-MB 2008
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Childhood Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia, children, adolescents, L-asparaginase, methotrexate
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Methotrexate; Cranial Irradiation; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Cranial irradiation (Active Comparator): Consolidation therapy with cranial irradiation in intermediate risk group patients
  Interventions: Radiation: Cranial irradiation
- Additional TIT (Experimental): Consolidation therapy with additional triple intrathecal therapy (N6) and without cranial irradiation in intermediate risk group patients
  Interventions: Drug: Triple intrathecal therapy
- MTX 2,000 mg/m2 (Experimental): Consolidation therapy with High-dose Methotrexate 2,000 mg/m2/24 h i.v. biweekly in intermediate risk group patients
  Interventions: Drug: High-dose Methotrexate
- MTX 30 mg/m2 (Active Comparator): Consolidation therapy with Low-dose Methotrexate 30 mg/m2 i.m. weekly in intermediate risk group patients
  Interventions: Drug: Low-dose Methotrexate
- PEG-asp 1,000 U/m2 (Experimental): Consolidation therapy with PEG-L-asparaginase cons 1,000 U/m2 biweekly in standard risk group patients
  Interventions: Drug: PEG-L-asparaginase cons
- L-asp 5,000 U/m2 (Active Comparator): Consolidation therapy with E.coli L-asparaginase 5,000 U/m2 weekly in standard risk group patients
  Interventions: Drug: E.coli L-asparaginase
- PEG-DNR+ (Active Comparator): Induction therapy without PEG-L-asparaginase and with Daunorubicin 45 mg/m2 in standard and intermediate risk group patients
  Interventions: Drug: Daunorubicin
- PEG+DNR+ (Experimental): Induction therapy with PEG-L-asparaginase ind (1,000 U/m2 on day 3 of therapy)and daunorubicin 45 mg/m2 in standard and intermediate risk group patients
  Interventions: Drug: PEG-L-asparaginase ind; Drug: Daunorubicin
- PEG+DNR- (Experimental): Induction therapy with PEG-L-asparaginase ind (1,000 U/m2 on day 3 of therapy) without daunorubicin on day 8 in standard risk group patients
  Interventions: Drug: PEG-L-asparaginase ind

INTERVENTIONS:
Drug: PEG-L-asparaginase ind — 1,000 U/m2 on day 3 of induction therapy, intravenously, in 200 ml of saline, during 1 hour
  Arms: PEG+DNR+; PEG+DNR-
Drug: PEG-L-asparaginase cons — 1,000 U/m2 intravenously, in 200 ml of saline, during 1 hour, 24 hours after methotrexate on weeks 7, 9, and 11 - days 44, 58, and 72 (phase S1), weeks 15, 17, and 19 - days 100, 114, 128 (phase S2), weeks 23, 25, and 27 - days 156, 170, 184 (phase S3).
  Arms: PEG-asp 1,000 U/m2
Drug: E.coli L-asparaginase — E.coli L-asparaginase (asparaginase medac) 5,000 U/m2 intramuscularly weekly, 24 hours after methotrexate dose, from week 7 to week 12 - days 44, 51, 58. 65, 72, 79 (phase S1), from week 15 to week 20 - days 100, 107, 114, 121, 128, 135 (phase S2), from week 23 to week 28 - days 156, 163, 170, 177, 184, 191 (phase S3).
  Other Names: Asparaginase Medac
  Arms: L-asp 5,000 U/m2
Drug: High-dose Methotrexate — 2,000 mg/m2 per 24 hours is given at days 43, 57, and 71 (weeks 7, 9, and 11). 1/5 of the total dose is given as slow intravenous bolus over 3-5 minutes. 4/5 of the total dose of methotrexate is injected as continuous 24 hours infusion.
  Arms: MTX 2,000 mg/m2
Drug: Low-dose Methotrexate — 30 mg/м2 is given intramuscularly 1 time weekly - days 43, 50, 57, 64, 71, and 78 (weeks 7, 8, 9, 10, 11, and 12).
  Arms: MTX 30 mg/m2
Drug: Triple intrathecal therapy — Intrathecal injection of 3 drugs is additionally given three times during phase S-2 (weeks 15, 17, and 19 - days 99, 113, and 127), and three times during phase S-3 (weeks 23, 25, and 27 - days 155, 169, and 183).
  Other Names: Methotrexate/Cytarabine/Prednisone i.th.
  Arms: Additional TIT
Radiation: Cranial irradiation — 12 Gy cranial irradiation is conducted at weeks 31-32 of the Protocol in patients >3 years of age
  Arms: Cranial irradiation
Drug: Daunorubicin — Daunorubicin at a dose of 45 mg/m2 i.v. for 6 hours on day 8 of induction therapy
  Arms: PEG+DNR+; PEG-DNR+

SUMMARY:
QUESTIONS AND OBJECTIVES OF ALL-MB-2008 STUDY

1. Whether the early PEG-asparaginase in induction will lead to the earlier achievement of remission, improvement of days 8 and 15 responses leading to an earlier reconstitution of bone marrow and immunocompetence, decrease of severe infections and early mortality rate?
2. Whether the use of PEG-asparaginase in induction will allow to avoid the anthracyclines in standard risk group patients and to reduce treatment myelotoxicity?
3. Whether the administration of 9 doses of PEG-asparaginase 1,000 U/m2 instead of 18 doses of E.coli L-asparaginase 5,000 U/m2 in standard risk patients will improve treatment outcome?
4. Whether the administrations of high dose methotrexate (2 g/m2 in 24 hours) during 1-st consolidation in intermediate risk patients will result in decrease of central nervous system relapse incidence and improvement of event-free and overall survival? Whether the increase of 6-mercaptopurine starting dose up to 50 mg/m2 in 1-st consolidation phase (instead of 25 mg/m2) will decrease in relapse risk, but would not be accompanied with enhanced toxicity?
5. Is it possible to completely avoid the cranial irradiation in intermediate risk patients? In some subgroup of intermediate risk patients? Is it enough to control neuroleukemia in these patients to introduce additional TIT in the consolidation phase of treatment? How will change the possible late effects in these patients according to the third arm of randomization?
6. Will the new risk group stratification to improve overall and event-free survival?

ELIGIBILITY:
Inclusion Criteria:

1. Age at diagnosis at 1 to 18 years.
2. The start of induction therapy within a time interval of study recruitment phase.
3. The diagnosis of ALL is to be proved by the morphological, cytochemical, and immunological analysis of tumor cells in bone marrow.
4. Informed consent of the parents (guardians) of the patient to be treated in one of the clinics included in this multicenter study.

Exclusion Criteria:

1. ALL is a second malignant tumor;
2. The disease is a relapse of previously misdiagnosed and, therefore, inadequately treated ALL;
3. There is severe concomitant disease, which significantly impedes chemotherapy protocol (such as multiple malformations, heart diseases, metabolic disorders, etc.);
4. There is a lack of important basic data needed for the exact adherence to the cytostatic therapy according to a specific protocol of chemotherapy (differential diagnosis of acute lymphoblastic/myeloid leukemia is not possible, stratification according to risk group is not possible);
5. The patient was treated before for a long time with cytotoxic drugs;
6. There were deviations in the treatment not covered by the protocol and/or not due to side effects of treatment and/or complications of the disease

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3000 (Estimated)
Dates: Start 2008-02 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 3 years, 5 years and 10 years after study start
overall survival | 3 years, 5 years and 10 years after study start
cumulative incidence of relapse | 3 years, 5 years and 10 years after study start

SECONDARY OUTCOMES:
early death rate | 3 years, 5 years and 10 years after study start
remission death rate | 3 years, 5 years and 10 years after study start

CONTACTS AND LOCATIONS:
Overall Officials: Alexander I. Karachunskiy, Professor, Principal Investigator — Research Institute of Pediatric Hematology, Oncology and Immunology
Locations (46):
- Belarus (3):
  - Republican Research and Practical Center of Radiation Medicine, Homyel
  - Republic Research and Practical Center of Pediatric Oncology and Hematology, Minsk
  - Mogilev Regional Children's Hospital, Mogilev
- Russia (42):
  - Arkhangelsk Regional Children's Hospital, Arkhangelsk
  - Regional Children's Hospital, Astrakhan
  - Moscow Regional Cancer Dispensary, Balashikha
  - Amur Regional Children's Hospital, Blagoveshchensk
  - Chelyabinsk Regional Children's Clinical Hospital, Chelyabinsk
  - Irkutsk Regional Children Clinical Hospital, Irkutsk
  - Regional Clinical Hospital, Ivanovo
  - Regional Children's Clinical Hospital, Khabarovsk
  - Kirov Research Institute of Hematology and Blood Transfusion, Kirov
  - Regional Children's Hospital, Krasnodar
  - Krasnoyarsk Territorial Clinical Children Hospital, Krasnoyarsk
  - Regional Children's Hospital, Kursk
  - Republic Children's Clinical Hospital, Makhachkala
  - Morozov Children's Clinical Hospital, Moscow
  - Research Institute of Pediatric Hematology, Oncology and Immunology named after Dmitry Rogachev, Moscow
  - Russian Children's Clinic Hospital, Moscow
  - Republic Children's Clinical Hospital, Nal'chik
  - District Children's Clinic Hospital, Nizhnevartovsk
  - Regional Children's Clinic Hospital, Nizhny Novgorod
  - Municipal Children's Clinic Hospital №4, Novokuznetsk
  - Novosibirsk Central District Hospital, Novosibirsk
  - Regional Clinical Oncology Dispensary, Orenburg
  - Perm Regional Children's Clinic Hospital, Perm
  - Regional Children's Hospital, Rostov-on-Don
  - Rostov Research Institute of Oncology, Rostov-on-Don
  - N. Dmitrieva Ryazan Regional Children's Hospital, Ryazan
  - Children's Municipal Hospital №1, Saint Petersburg
  - Municipal Hospital №31, Saint Petersburg
  - R. Gorbacheva Research Institute of Pediatric Hematology and Transfusiology; Pavlov State Medical University of Saint-Petersburg, Saint Petersburg
  - Children's Municipal Clinical Hospital №1, Samara
  - Profpathology and Hematology Clinic; Saratov State Medical University, Saratov
  - Regional Children's Clinical Hospital, Stavropol
  - Surgut Central District Clinical Hospital, Surgut
  - Tomsk Regional Clinical Hospital, Tomsk
  - Tula Regional Children's Hospital, Tula
  - Republic Children's Clinical Hospital, Ulan-Ude
  - Ulyanovsk Regional Children's Clinical Hospital, Ulyanovsk
  - Municipal Children's City Hospital, Territorial Children's Hematological Center, Vladivostok
  - Voronezh Regional Children Clinical Hospital №1, Voronezh
  - Republic Hospital №1 - National Medicine Centre, Yakutsk
  - Regional Children's Clinical Hospital, Yaroslavl
  - Regional Children's Clinical Hospital № 1, Yekaterinburg
- Research Institute of Hematology and Blood Transfusion, Tashkent, Uzbekistan

REFERENCES:
- See also: Study web-site — http://www.mbstudy.net